CLINICAL TRIAL: NCT05063448
Title: DadSpace: Increasing Community Support Resources for Perinatal Fathers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other)
Responsible Party: Principal Investigator, Julie Rieker, Department Head and Professor, Colorado State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1754
Record Dates: First submitted 2021-09-08; First posted 2021-10-01 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Paternal Behavior; Father-Child Relations; Family Relations
Keywords: Perinatal

STUDY DESIGN:
Intervention Model Description: Perinatal father support primary intervention is small group mentoring program (with pre/post test data) run by educators at The Women's Clinic (TWC). Participants who sign up for the program early enough will be provided surveys approximately 1 month prior to the intervention start to provide a non-randomized wait-list comparison. Participants will additionally have access to follow-up daddy/baby drop-in groups and a podcast series and may be provided satisfaction surveys for both.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DadSpace Intervention (Experimental): Participants will take part in a 12-hour educational discussion-based mentoring program intervention over 8 weeks. The intervention will be facilitated by a trained father facilitator and will include education and support on topics relevant to perinatal fathers. Topics include father identity, stress management, infant development, co-parenting, masculinity and caregiving, healthy communication, and work-life balance. Participants will additionally have access to a brief educational podcast series on related topics. Participants will also be invited to monthly follow-up daddy/baby drop-in groups.
  Interventions: Behavioral: DadSpace

INTERVENTIONS:
Behavioral: DadSpace — A group educational support and mentoring program for perinatal fathers.

SUMMARY:
The project is aimed at meeting the support needs of community fathers who are expecting a baby or who have recently had a baby. This work is being conducted in conjunction with community partners through The Women's Clinic of Northern Colorado (WCNC). Researchers and WCNC staff will work together to develop and implement programs for prenatal and postpartum fathers. Participants will be invited to a group mentoring program and also will be provided access to supplementary educational podcasts focused on topics relevant to prenatal and postpartum fathers. The investigators are seeking to understand what participants like and don't like about the program and how participation in the program affects participants' stress, well-being, and parenting.

DETAILED DESCRIPTION:
The investigators are building on previous work to identify opportunities to meet the needs of perinatal fathers. The term perinatal encompasses the time leading up to and immediately following the birth of a child. Father involvement in child rearing is beneficial to mothers and children, but fathers are routinely overlooked by available support opportunities at the transition to parenthood. This pilot project seeks to apply research evidence and best practices to address the disparity in socioemotional community support and education programs serving perinatal fathers. In a previous pilot study, the investigators learned from fathers participating in focus groups that participants were interested in opportunities to connect with other fathers in the same life stage to talk about personal experiences and learn from each other. The investigators also learned that fathers worry about meeting varied role expectations, that available resources tend to overlook the unique experiences of fathers, and that it can be challenging to find quality information in a digital world saturated with conflicting information about parenting. This project seeks to address these primary issues through community-based, father-centric support and educational programs. WCNC education staff will facilitate a discussion-based group mentoring program for fathers who are expecting or recently had a baby. This program seeks to increase connection with other fathers, reduce stress related to parenting a baby, and increase parenting confidence. The investigators plan to evaluate the feasibility of the program through satisfaction surveys and other measures of the program's implementation. The investigators also plan to evaluate the effectiveness of the program by providing participants with surveys asking about their well-being, knowledge, confidence in parenting, and their satisfaction with their social networks. The investigators are additionally developing educational podcasts focused on topics relevant to prenatal and postpartum fathers, which will be evaluated as a supplementary component to the mentoring program. Research objectives are the following: Study 1, Objective 1 (Primary): The investigators seek to determine the feasibility and acceptability of a program targeting perinatal fathers offered in a community clinic setting. Study 1, Objective 2 (Primary): Examine whether participating in a discussion-based group mentoring program increases the likelihood of positive short-term outcomes for fathers. Study 1 Objective 3 (Secondary): Identify whether listening to brief, targeted educational podcasts predicts increased positive outcomes for fathers over and above the mentoring group alone. Study 2 Objective 1 (Primary): Identify whether participants who listen to brief, targeted educational podcasts find the podcasts satisfactory and acceptable as a method of gaining information about perinatal fatherhood.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be expecting a baby or have a baby less than one year of age and planning to take the DadSpace mentoring program.

Exclusion Criteria:

* Non-English speaking

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — If participant identifies as male or as a father, whether or not participant is biologically male, participant may be included in the study.
Enrollment: 20 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Braungart-Rieker, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DadSpace Intervention
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.21 (4.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19
Marital Status [Count of Participants; unit: Participants]
  Married | 18
  Single never married | 1
  Divorced | 0
  Widowed | 0
Household Income [Count of Participants; unit: Participants]
  $20,000-39,999 | 1
  $40,000-59,999 | 2
  $60,000-84,999 | 1
  $85,000+ | 15
Birth Status: Prenatal, Postpartum [Count of Participants; unit: Participants]
  Prenatal, expecting baby | 12
  Postpartum, baby has been born | 7
Residential Status: Reside or Not Reside with Infant [Count of Participants; unit: Participants]
  Resides in home with infant | 6
  Does not reside in home with infant | 1
  N/A (baby not born) | 12
Additional Children: Yes, No [Count of Participants; unit: Participants]
  Also has older children | 1
  Does not also have older children | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Knowledge of Infant Development Inventory
Description: This 19-item abbreviated version of the inventory assesses accurate knowledge of infant development. The first 11 items are rated as true or false and include questions such as "Babies may cry for 20-30 minutes at a time, no matter how much you try to comfort them" and "Some parents do not bond until their baby starts to smile and look at them." An additional 6 items ask parents to rate whether they think babies can do something at the age listed in the item or whether the developmental task (e.g., "Six-month-olds know what 'no' means.") occurs in younger or older children. Two additional items ask respondents to choose the best way to respond to potentially stressful infant behaviors (breaking things and fussing at night). Item responses are scored as correct or incorrect with percent correct as the final measure.
Time Frame: Every 4 weeks up to 16 weeks, including pre-intervention, mid-intervention, post-intervention, and follow-up
Population: Participants who participated in baseline and posttest surveys.
Measure: Mean (Standard Deviation); unit: Percent correct
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 18
Percent correct
  Baseline | 77.78 (10.3)
  Mid-intervention | 81.87 (6.56)
  Posttest | 67.25 (13.70)
  Follow-up: number analyzed (Participants) | 15
  Follow-up | 78.95 (11.43)

2. Primary Outcome: Change in Self-Perceptions of the Parental Role-Competence Scale
Description: A 6-item measure of feelings of efficacy/competence in the parental role. Items are weighted on a range from 1 to 4, with higher scores indicating higher confidence in the parental role, a better outcome. Scores are totaled with a possible range from 4 to 24.
Time Frame: Every 4 weeks up to 16 weeks, including pre-intervention, mid-intervention, post-intervention, and follow-up
Population: DadSpace participants who completed the posttest survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 18
score on a scale
  Baseline | 17.18 (3.57)
  Mid-intervention | 18.39 (3.24)
  Posttest | 18.89 (3.12)
  Follow-up: number analyzed (Participants) | 15
  Follow-up | 19.33 (3.70)
Statistical Analysis 1: Comparison: DadSpace Intervention; Reliable change indices compare participants to themselves from Time 1 (baseline) and Time 3 (post-intervention). Reliable change indices measure whether the score change of individual participants is more than would be expected based on measurement error alone. Reliable change results are presented as number of participants who fell outside of the reliable change confidence interval in each direction indicating reliable increases or decreases in score; Test type: Other — Reliable change is calculated by multiplying the standard deviation of the measure by Cronbach's alpha reliability to determine the standard error of the measure. The standard error of the measure is multiplied by 1.96 to calculate a confidence interval around the line of no change, when the slope of pre-test to post-test = 1. Using time 3 parameters, the reliable change index for this scale was ±2.47. Cases that fall outside of the confidence interval are considered to show reliable change; Slope = 1.00, 95% CI 2-sided [-1.47 to 3.47] — Five cases fell outside of the upper confidence interval
Statistical Analysis 2: Comparison: DadSpace Intervention; Paired samples t-test was used to compare group average pretest (time 1) and posttest (time 3) scores of self-perceptions of the parental role, a measure of parenting confidence; Test type: Superiority; p = 0.022, t-test, 2 sided — This is not adjusted for multiple comparisons. A priori alpha is set at 95% with two tails; t = 2.547, df = 16. N at time 3 = 18

3. Primary Outcome: Change in Social Network Questionnaire-Satisfaction Scale
Description: 7 yes/no items on satisfaction with the support received from one's social network. More "yes" answers indicates lower satisfaction with the social network, a worse outcome. Scores are reverse-scored and totaled with a possible range from 0 to 7 so that higher scores indicate more satisfaction.
Time Frame: Every 4 weeks up to 16 weeks, including pre-intervention, mid-intervention, post-intervention, and follow-up
Population: DadSpace participants who completed surveys at any of the time-points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 18
score on a scale
  Baseline | 4.56 (2.23)
  Mid-intervention | 4.72 (2.32)
  Posttest | 4.67 (2.38)
  Follow-up: number analyzed (Participants) | 15
  Follow-up | 4.80 (2.37)
Statistical Analysis 1: Comparison: DadSpace Intervention; [analysis description as in outcome 2, analysis 1]; Test type: Other — Reliable change is calculated by multiplying the standard deviation of the measure by Cronbach's alpha reliability to determine the standard error of the measure. The standard error of the measure is multiplied by 1.96 to calculate a confidence interval around the line of no change, when the slope of pre-test to post-test = 1. Using time 3 parameters, the reliable change index for this scale was ±1.84. Cases that fall outside of the confidence interval are considered to show reliable change; Slope = 1.00, 95% CI 2-sided [-0.84 to 2.84] — Three cases fell outside of the upper confidence interval

4. Primary Outcome: Change in Role Conflict Scale
Description: 2 subscales that assess work conflict with family life, family life conflict with work, and work-family balance. Item values range from 1 to 6. Higher scores indicate a worse outcome. Scores are totaled with a possible range of 8 to 48.
Time Frame: Every 4 weeks up to 16 weeks, including pre-intervention, mid-intervention, post-intervention, and follow-up
Population: Participants who completed surveys at any time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 18
score on a scale
  Baseline | 21.50 (7.22)
  Mid-intervention | 21.00 (7.98)
  Posttest | 22.22 (7.47)
  Follow-up: number analyzed (Participants) | 15
  Follow-up | 20.80 (8.81)
Statistical Analysis 1: Comparison: DadSpace Intervention; [analysis description as in outcome 2, analysis 1]; Test type: Other — Reliable change is calculated by multiplying the standard deviation of the measure by Cronbach's alpha reliability to determine the standard error of the measure. The standard error of the measure is multiplied by 1.96 to calculate a confidence interval around the line of no change, when the slope of pre-test to post-test = 1. Using time 3 parameters, the reliable change index for this scale was ±5.97. Cases that fall outside of the confidence interval are considered to show reliable change; Two cases demonstrated reliable and one case demonstrated a reliable increase in work-family role conflict at posttest; Slope = 1.00, 95% CI 2-sided [-4.97 to 6.97] — Two cases fell outside of the upper confidence interval and one case fell outside of the lower confidence interval

5. Primary Outcome: Change in Perceived Stress Scale
Description: 10 items related to anxiety, stress, and coping with upsets. Items values range from 0 to 4 with higher scores indicating higher perceived stress, a worse outcome. Scores are totaled with a possible range from 0 to 40.
Time Frame: Every 4 weeks up to 16 weeks, including pre-intervention, mid-intervention, post-intervention, and follow-up
Population: DadSpace participants who completed surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 18
score on a scale
  Baseline | 16.66 (5.48)
  Mid-intervention | 15.61 (6.12)
  Posttest | 16.50 (7.21)
  Follow-up: number analyzed (Participants) | 15
  Follow-up | 17.00 (5.84)
Statistical Analysis 1: Comparison: DadSpace Intervention; [analysis description as in outcome 2, analysis 1]; Test type: Other — Reliable change is calculated by multiplying the standard deviation of the measure by Cronbach's alpha reliability to determine the standard error of the measure. The standard error of the measure is multiplied by 1.96 to calculate a confidence interval around the line of no change, when the slope of pre-test to post-test = 1. Using time 3 parameters, the reliable change index for this scale was ±4.78; Slope = 1.00, 95% CI 2-sided [-3.78 to 5.78] — Three cases fell below the confidence interval and two cases fell above the confidence interval

6. Primary Outcome: Change in Edinburgh Postnatal Depression Scale
Description: 10 items that measure core features of postnatal depression. Item values range from 0 to 3 with a higher score indicating higher depressive symptoms, a worse outcome. Scores are totaled with a possible range from 0 - 30.
Time Frame: Every 4 weeks up to 16 weeks, including pre-intervention, mid-intervention, post-intervention, and follow-up
Population: DadSpace participants who completed surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 18
score on a scale
  Baseline | 7.17 (6.19)
  Mid-intervention | 6.39 (5.45)
  Posttest | 7.22 (5.82)
  Follow-up: number analyzed (Participants) | 15
  Follow-up | 7.67 (5.07)
Statistical Analysis 1: Comparison: DadSpace Intervention; [analysis description as in outcome 2, analysis 1]; Test type: Other — Reliable change is calculated by multiplying the standard deviation of the measure by Cronbach's alpha reliability to determine the standard error of the measure. The standard error of the measure is multiplied by 1.96 to calculate a confidence interval around the line of no change, when the slope of pre-test to post-test = 1. Using time 3 parameters, the reliable change index for this scale was ±3.37. Cases that fall outside of the confidence interval are considered to show reliable change; Slope = 1.00, 95% CI 2-sided [-2.27 to 4.37] — Three cases fell below the lower confidence interval and two cases fell above the upper confidence interval

7. Primary Outcome: Change in Spielberger State Anxiety Scale (Short Form)
Description: 10 items assessing feelings of upset and anxiety versus contentment at the present time. Item values range from 1 to 4 with a higher score indicating higher state anxiety, a worse outcome. Scores are totaled with a total possible range from 6 to 24.
Time Frame: Every 4 weeks up to 16 weeks, including pre-intervention, mid-intervention, post-intervention, and follow-up
Population: DadSpace participants who completed surveys at any timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 18
score on a scale
  Baseline | 11.33 (4.52)
  Mid-intervention | 10.89 (4.44)
  Posttest | 11.94 (3.99)
  Follow-up: number analyzed (Participants) | 15
  Follow-up | 11.47 (4.21)
Statistical Analysis 1: Comparison: DadSpace Intervention; [analysis description as in outcome 2, analysis 1]; Test type: Other — Reliable change is calculated by multiplying the standard deviation of the measure by Cronbach's alpha reliability to determine the standard error of the measure. The standard error of the measure is multiplied by 1.96 to calculate a confidence interval around the line of no change, when the slope of pre-test to post-test = 1. Using time 3 parameters, the reliable change index for this scale was ±2.80. Cases that fall outside of the confidence interval are considered to show reliable change; Slope = 1.00, 95% CI 2-sided [-1.80 to 3.80] — Two cases fell below the lower confidence interval and two cases fell above the upper confidence interval

8. Primary Outcome: Change in Coparenting Relationship Scale - Brief
Description: 13 items assessing coparent collaboration versus conflict related to child rearing. Items values range from 0 to 6 with higher scores indicating a better coparenting relationship. Items are totaled with a possible range from 0 - 72.
Time Frame: Every 4 weeks up to 16 weeks, including pre-intervention, mid-intervention, post-intervention, and follow-up
Population: Participants who completed surveys at any time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 18
score on a scale
  Baseline | 51.83 (5.51)
  Mid-intervention | 51.94 (7.95)
  Posttest | 51.00 (8.19)
  Follow-up: number analyzed (Participants) | 15
  Follow-up | 51.00 (7.67)

9. Secondary Outcome: Change in Pearlin Mastery Scale
Description: 7-item measure of general self-efficacy versus helplessness. Item values range from 1 to 6 with higher scores indicating worse self-efficacy. Scores are totaled with a total possible range from 6 to 42.
Time Frame: Every 4 weeks up to 16 weeks, including pre-intervention, mid-intervention, post-intervention, and follow-up
Population: DadSpace participants who completed surveys at any time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 18
score on a scale
  Baseline | 33.83 (5.96)
  Mid-intervention | 33.11 (6.72)
  Posttest | 31.94 (7.71)
  Follow-up: number analyzed (Participants) | 15
  Follow-up | 30.87 (7.99)
Statistical Analysis 1: Comparison: DadSpace Intervention; [analysis description as in outcome 2, analysis 1]; Test type: Other — Reliable change is calculated by multiplying the standard deviation of the measure by Cronbach's alpha reliability to determine the standard error of the measure. The standard error of the measure is multiplied by 1.96 to calculate a confidence interval around the line of no change, when the slope of pre-test to post-test = 1. Using time 3 parameters, the reliable change index for this scale was ±4.03. Cases that fall outside of the confidence interval are considered to show reliable change; Slope = 1.00, 95% CI 2-sided [-3.03 to 5.03] — One case fell outside of the upper confidence interval, while 5 participants fell below the lower confidence interval

10. Secondary Outcome: Change in Paternal Postnatal Attachment Scale
Description: Assesses fathers' positive feelings versus lack of enjoyment with the baby. Item values have been revised from the original scale to range from 1 to 6 with higher scores indicating more positive feelings toward the baby. Scores are totaled with a possible range from 19 to 114.
Time Frame: Every 4 weeks up to 16 weeks, including pre-intervention, mid-intervention, post-intervention, and follow-up
Population: Participants who completed surveys and whose babies have been born by the selected time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 10
score on a scale
  Baseline: number analyzed (Participants) | 7
  Baseline | 101.20 (11.86)
  Mid-intervention: number analyzed (Participants) | 7
  Mid-intervention | 92.53 (18.89)
  Posttest: number analyzed (Participants) | 9
  Posttest | 93.44 (16.44)
  Follow-up | 92.50 (15.64)

11. Other Pre Specified Outcome: Attendance
Description: Number of total sessions attended by participants (dosage)
Time Frame: Measured across the 8 weeks of intervention delivery with one session offered per week.
Population: Perinatal fathers who participated in the DadSpace program.
Measure: Mean (Standard Deviation); unit: total number of sessions attended
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 19
total number of sessions attended | 6.56 (1.72)

12. Other Pre Specified Outcome: Facilitator Fidelity to Protocol
Description: A checklist of intervention items completed by the facilitator to identify adherence to the intervention protocol.
Time Frame: Measured across the 8 weeks of intervention delivery
Population: Average fidelity across the two facilitators of the program
Measure: Mean (Full Range); unit: percentage of manual items covered
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 2
percentage of manual items covered | 92 [79 to 100]

13. Other Pre Specified Outcome: Helpfulness of Information Sources
Description: Fathers report on how helpful they found the provided resources (e.g., handouts) on a scale from 1 to 4 with a higher score indicating a higher degree of helpfulness, a better outcome.
Time Frame: Measured at posttest, 8 weeks after pretest.
Population: Participants who attended at least two sessions of the program and completed the posttest survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 18
score on a scale | 3.53 (0.51)

14. Other Pre Specified Outcome: Participant Engagement
Description: Facilitator ratings of participants' active participation and evidence that fathers have been trying out skills covered in classes. Engagement was measured by totaling scores from two items. Item one asked facilitator's to rate how active participants were in participating in class measured on a scale from 0 (passive) to 5 (active). Item two asked facilitators to rate the degree to which they have observed the participants trying out the skills they are learning in class on a scale from 0 (not at all) to 3 (yes, quite a lot). After summing scores for the two items, engagement has a possible range of 0-8. Higher scores indicate more engagement, a better outcome.Total scores were averaged to produce a single score of engagement across all weekly sessions and cohorts.
Time Frame: Measured after each of 8 weekly sessions. Scores for each week were averaged to produce a total score of engagement for all participants.
Population: Facilitators reported an overall score for all participants in each session. Scores were averaged across weeks and cohorts to produce an overall engagement score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 19
units on a scale | 5.83 (2.08)

15. Other Pre Specified Outcome: Support Group Social Exchange Scale
Description: The 27-item Support Group Social Exchange Scale assesses various types of social exchanges that can occur in support group dynamics, including experiential knowledge, emotional support, humor, and unwanted behavior. We removed three of the five items asking about humor, reducing the number of items to 24. Items statements (e.g., "I shared my personal problems with group members") are rated from 0 (never) to 6 (always). Three items ask participants to rate the number of times they interacted with other participants outside of group meetings, such as by doing favors for and socializing with each other, with ordinal response categories ranging from 0 (0 times) to 4 (10 or more times). Item scores are summed to produce a total score for each participant with a possible range from 0 to 156. Higher scores indicate a more positive perception of group social dynamics, a better outcome.
Time Frame: Immediately after the intervention
Population: Perinatal fathers who completed at least two weeks of the program and completed the posttest survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 18
score on a scale | 118.94 (16.71)

16. Other Pre Specified Outcome: Satisfaction With DadSpace Program
Description: Fathers rate their overall satisfaction with the utility of each of the eight sessions on a scale from 0 to 10 with higher scores indicating more satisfaction. Scores are averaged for an average satisfaction score.
Time Frame: Immediately after the end of the intervention
Population: Participants who completed at least two weeks of the DadSpace program and completed the posttest survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 18
score on a scale | 8.10 (2.03)

17. Other Pre Specified Outcome: Workshop Environment Scale
Description: The Workshop Environment Scale provides a measure of group dynamics and facilitator alliance. Items were adapted to fit the specific program and reduced to 10 questions scaled from 1 (strongly disagree) to 4 (strongly agree), with higher scores indicating more positive perceptions of the workshop environment, a better outcome. Item scores were summed to produce a total score with a possible range of 4 to 40.
Time Frame: Participants completed the workshop environment scale at posttest (time 3).
Population: Perinatal fathers who completed at least two weeks of the program and completed the posttest survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DadSpace Intervention
Number analyzed (Participants) | 18
score on a scale | 34.88 (4.11)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during study surveys at mid-intervention (4 weeks), posttest (8 weeks), and follow-up (12 weeks)
Arm/Group | DadSpace Intervention
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 1/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DadSpace Intervention (N=19)
Thoughts of self-harm with no intervention needed (Psychiatric disorders) | 1 (1) — Participant endorsed "Yes, quite often" for "The thought of harming myself has occurred to me" on the Edinburgh postnatal depression scale at the mid-intervention survey. Participant indicated no immediate risk of harm and was provided resources.

LIMITATIONS AND CAVEATS:
We were not able to recruit sufficient participants to have a wait-list comparison group, as originally intended. All outcomes should therefore be considered only exploratory in nature and not conclusive of intervention effectiveness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/48/NCT05063448/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT05063448/SAP_001.pdf